CLINICAL TRIAL: NCT05009654
Title: Carnitine Supplementation and Skeletal Muscle Function in Aging
Brief Title: The Effect of Leucine on Carnitine Transport to Skeletal Muscle
Acronym: ROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCN_ROL; 2014/15/B/NZ7/00893 (Other Grant/Funding Number: National Science Centre)
Record Dates: First submitted 2021-08-05; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Carnitine; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carnitine + leucine (Experimental): 1000 mg L-carnitine with 3000 mg L-leucine per day for 24 weeks
  Interventions: Dietary Supplement: L-carnitine; Dietary Supplement: L-leucine
- leucine (Placebo Comparator): 4000 mg L-leucine per day for 24 weeks
  Interventions: Dietary Supplement: L-leucine

INTERVENTIONS:
Dietary Supplement: L-carnitine
  Other Names: L-carnitine-L-tartrate
  Arms: carnitine + leucine
Dietary Supplement: L-leucine

SUMMARY:
The primary aim of the current research project is to explore whether leucine stimulates carnitine transport, and thus affecting muscle carnitine content.

A secondary aim of this project is to investigate the effect of carnitine with leucine supplementation on muscle strength and body composition.

ELIGIBILITY:
Inclusion Criteria:

* must be able to swallow tablets

Exclusion Criteria:

* cardiovascular disease
* liver disease
* kidney disease
* neuromuscular disease
* gastrointestinal disorders (including stomach ulcers and erosions)
* diabetes
* other severe chronic diseases

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Muscle Carnitine Concentration using UPLC-MS/MS | 24 weeks
  vastus lateralis muscle biopsy taken before and after the supplementation procedure (~20 cm proximal to the knee joint using a thin biopsy needle); carnitine concentration determined using ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) method

SECONDARY OUTCOMES:
Muscle Strength using Biodex System 4 Pro dynamometer | 24 weeks
  Peak torque measured by performing maximum voluntary contractions during isometric knee extension and flexion. The test performed in concentric-concentric mode consisting maximum 4-s knee extensor isometric contraction and maximum 4-s knee flexor isometric contraction, separated by 20-s recovery, repeated three times. Muscle isokinetic strength assessed in 5 repetitions of flexion and extension at a speed of 60°/s. Muscle endurance assessed in 10 repetitions at 300°/s determine the ability of the muscle to maintain the work. Strength testing performed on the Biodex System 4 Pro dynamometer.
Body Composition: Body Fat Mass, Fat Free Mass, and Skeletal Muscle Mass using a bioelectrical impedance analyzer (InBody720). | 24 weeks
  The InBody720 measures impedance of five segments of the body (each arm, each leg, trunk) at frequencies of 1, 5, 50, 250, 500, and 1000 kHz through the 8-polar tactile-electrode. Based on the impedance, body fat mass, fat free mass, and skeletal muscle mass are calculated.